CLINICAL TRIAL: NCT01624025
Title: A Comparative Study of Salvage Treatment With Combination of Docetaxel and Epirubicin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0222
Record Dates: First submitted 2012-06-12; First posted 2012-06-20 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Advanced Gastric Cancer
Keywords: AGC, second-line, docetaxel, epirubicin
MeSH Terms: interventions — Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HER2 positive (Experimental): Both the patients with HER2 (+) and HER2 (-) patients will be treated with the same regimen.(Docetaxel 60 mg/m2, epirubicin 60 mg/m2, q3wks)
  Interventions: Other: Docetaxel 60 mg/m2, epirubicin 60 mg/m2, q3wks
- HER2 negative (Active Comparator): Both the patients with HER2 (+) and HER2 (-) patients will be treated with the same regimen.
  (Docetaxel 60 mg/m2, epirubicin 60 mg/m2, q3wks)
  Interventions: Other: Docetaxel 60 mg/m2, epirubicin 60 mg/m2, q3wks

INTERVENTIONS:
Other: Docetaxel 60 mg/m2, epirubicin 60 mg/m2, q3wks — Both the patients with HER2 (+) and HER2 (-) patients will be treated with the same regimen.

SUMMARY:
A salvage treatment with combination of docetaxel and epirubicin in patients with unresectable, metastatic gastric cancer after fluoropyrimidine failure : A HER2 status-based study

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic, or recurrent AGC
2. Previous use of fluoropyrimidine as palliative chemotherapy. Concurrent use of platinum is permitted. Patient with recurred disease within 6 months after the end of adjuvant therapy can participate to this trial.
3. Documented HER2 expression status.
4. Radiologically proven progression of disease.
5. Age > 20 years
6. ECOG PS 0 - 2
7. Life expectancy more than 3 months
8. Adequate organ function for treatment including liver, kidney and bone marrow (absolute neutrophil count (ANC) ≥ 1,500/ul, platelets ≥ 100,000/ul, AST/ALT ≤ 2.5 x ULN, ≤ 5.0 x ULN if liver involvement, Total serum bilirubin ≤ 2.0 mg/dL)
9. Written informed consent

Exclusion Criteria:

1. Prior administration of taxane or anthracycline as palliative chemotherapy. If those agents were used as adjuvant or neoadjuvant aim, at least 6 months should be passed.
2. Uncontrolled medical comorbidities Congestive heart failure (NYHA class III or IV) Recent (within 6 months) unstable angina or myocardial infarct Clinically significant cardiac arrhythmia LVEF < 45% Liver cirrhosis (Child-Pugh class B or C) Interstitial pneumonia Psychiatric illness/social situations that would limit compliance with study requirements
3. Active CNS metastasis not controllable with radiation or steroid
4. Concurrent administration of systemic chemotherapy or radiotherapy. Palliative radiotherapy for pain control more than 2 weeks ago is acceptable.
5. Pregnant or lactating women.
6. Peripheral neuropathy G3~4.
7. Metachronous malignancy other than adequately treated CIN of uterine cervix, basal cell or squamous cell carcinoma of the skin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
disease control rate according to the RECIST v1.1 | at 6~8 weeks later after the first evaluation
  The primary outcome of the current study is the disease control according to the HER2 status. That is, the % of the patients who maintains at least stable disease by RECIST v1.1 at the time of the second tumor evaluation which will be taken at 6~8 weeks later after the first evaluation. The comparison will be done by Pearsons's chi-square test.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea